CLINICAL TRIAL: NCT06567938
Title: Intravascular Ultrasound-Guided or Angiography-Guided Percutaneous Coronary Intervention in Patients With Chronic Kidney Disease: The IVUS-CKD Trial
Brief Title: Intravascular Ultrasound-Guided PCI in Patients With Chronic Kidney Disease
Acronym: IVUS-CKD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HXIIT2024007
Record Dates: First submitted 2024-07-10; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-06

CONDITIONS: Coronary Artery Disease; Chronic Kidney Diseases
Keywords: Coronary Artery Disease; Chronic Kidney Disease; Percutaneous Coronary Intervention; Intravascular Ultrasound; Randomized Trial
MeSH Terms: conditions — Coronary Artery Disease; Renal Insufficiency, Chronic | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVUS-guidance PCI (Experimental): In the IVUS-guidance group, the optimal stent deployment criteria for non-left main lesion will include the following: : (1) the minimal lumen area (MLA) in the stented segment > 5.0 mm^2 or > 90% of the MLA at the distal reference segments, (2) plaque burden 5 mm proximal or distal to the stent edge is < 55%, and (3) absence of medial dissection over 3 mm in length. In the setting of a two-stent approach for distal left main bifurcation lesions, the optimal stent deployment criteria are an absolute minimal stent area (MSA) greater than 8 mm^2 for the left main, greater than 7 mm^2 for carina, greater than 6 mm^2 for the ostial or proximal left anterior descending artery, and greater than 5 mm^2 for the ostial or proximal left circumflex artery. For left main lesion treated with single-stent technique, the criteria are greater than 7mm^2 for distal and greater than 8mm^2 for proximal. Further treatment will be required if the criteria are not met.
  Interventions: Procedure: Percutaneous coronary intervention
- Angiography-guidance PCI (Active Comparator): Angiographic success is defined as thrombolysis in myocardial infarction (TIMI) flow grade 3, and residual stenosis < 20%.
  Interventions: Procedure: Percutaneous coronary intervention

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — PCI with DES implantation
  Other Names: PCI

SUMMARY:
The IVUS-CKD study is a prospective, randomized controlled, multicenter trial to determine whether the intravascular ultrasound (IVUS)-guided percutaneous coronary intervention is superior to the angiography-guidance in chronic kidney disease (CKD) patients with respect to target vessel failure (TVF) at 12 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

* CKD patients with eGFR<60 mL/min/1.73 m^2
* De novo coronary lesion suitable for second-generation metallic drug-eluting stent placement and IVUS imaging
* Signed written informed consent

Exclusion Criteria:

* Onset of STEMI within 24 hours or emergent angiography
* Pregnant or childbearing women
* Co-morbidity with an estimated life expectancy of < 1 year
* LVEF ≤ 30%
* Cardiogenic shock or hemodynamic instability
* Severe hepatic dysfunction, defined as ALT or AST more than 5 times the ULN
* PCI within the previous 12 months
* Target lesion of stent thrombosis or in-stent restenosis
* Any planned non-cardiac surgery within 12 months
* Inability to follow the protocol and comply with follow-up requirements or any other reason that the investigator feels would place the patient at increased risk
* Current enrolment in other clinical trials
* Contraindication to anti-platelet agents
* History of intracranial or gastrointestinal bleeding requiring transfusion or surgical intervention for control (excluding hemorrhoid)
* Chronic total occlusion lesion with unsuccessful guidewire crossing
* Current intake of nephrotoxic medications (e.g., nonsteroidal anti-inflammatory drugs except acetylsalicylic acid, phenylbutazone, aminoglycosides, amphotericin B, polymyxin, platinum complexes)
* Immune-related kidney disease or on hormone therapy (e.g. lupus nephritis, IgA nephropathy)
* Planned exposure to contrast within 72 h after the procedure, intravascular administration of contrast within the previous 5 days
* Intake of anticoagulants
* Hemoglobin <60 g/L
* Severe valvular disease or valvular disease likely to require surgery or percutaneous valve replacement during the trial
* Patients allergic to metals or contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1528 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Target vessel failure (TVF), including cardiac death, target vessel myocardial infarction (MI), or clinically driven target vessel revascularization (TVR) | 12 months
  The difference in TVF will be calculated from 0 month to 12 months between IVUS- and Angiography-guidance groups.

SECONDARY OUTCOMES:
Hierarchical composite of target vessel failure | 12 months
  Hierarchical composite of cardiac death, target vessel MI, or clinically driven target vessel revascularization after randomization analyzed by win ratio method.
30-day cardiorenal endpoint | 30 days
  A composite of contrast-associated acute kidney injury (CA-AKI), requiring specific treatment for acute renal failure, persistent decline in eGFR, MI, or all-cause death.
Target vessel failure excluding periprocedural MI | 12 months
  The difference will be calculated from 0 month to 12 months between IVUS- and Angiography guidance groups.
Cardiac death | 12 months
  Death that could not be attributed to a noncardiac etiology is considered cardiac death.
Target vessel MI | 12 months
Clinically driven target vessel revascularization | 12 months
  Any clinically driven repeat percutaneous intervention or surgical bypass of any segment of the target vessel including the target lesion.
Spontaneous MI | 12 months
Target lesion failure | 12 months
  A composite of cardiac death, target vessel related MI, or clinically driven target lesion revascularization.
Clinically driven target lesion revascularization | 12 months
Major adverse cardiovascular event | 12 months
  A composite of cardiac death, MI, definite stent thrombosis (ST), or clinically driven TVR

OTHER OUTCOMES:
Renal outcomes | 12 months
  A composite of requiring specific treatment for acute renal failure (continuous renal replacement therapy, or dialysis), chronic dialysis (peritoneal dialysis, or hemodialysis), persistent decline in eGFR, or renal death.
Annual change in eGFR from baseline | 12 months
  total slope
Clinically relevant bleeding | 12 months
  Bleeding Academic Research Consortium Definition for Bleeding types 2，3 or 5
Major bleeding | 12 months
  Bleeding Academic Research Consortium Definition for Bleeding types 3 or 5
All-cause death | 12 months
Definite or probable stent thrombus (ST) | 12 months
  ST was classified as definite, probable, or possible, according to the definitions provided by the Academic Research Consortium (ARC).
Procedure time | during PCI
  From first wire insertion to guide catheter removal.
Radiation exposure | during PCI
  From first wire insertion to guide catheter removal.
Total amount of contrast use | during PCI
  From first wire insertion to guide catheter removal.

CONTACTS AND LOCATIONS:
Overall Officials: Ning Guo, Principal Investigator — The First Affiliated of Xi'an Jiaotong University
Locations (1):
- The First Affiliated Hopital of Xi'an Jiaotong University, Xi'an, Shaanxi, China